CLINICAL TRIAL: NCT01415648
Title: Medico-economic Evaluation of Preoperative Cerebral Oximetry Monitoring During Carotid Endarterectomy.
Acronym: EMOCAR
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment time expired.
Sponsor: Nantes University Hospital (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: STIC/10/02; 2010-A01167-32 (Other: Afssaps)
Record Dates: First submitted 2011-07-11; First posted 2011-08-12 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Internal Carotid Stenosis
Keywords: with surgical indication; Cerebral oximetry; carotid endarterectomy; MRI; ischemic lesion; cost/effectiveness analysis; Neurocognitive Outcome; protein S-100B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- open NIRS (Experimental): continuous per operative cerebral oximetry monitoring (using INVOS™ cerebral oximeter) associated with hemodynamic optimisation algorithm (excluding norepinephrine) if cerebral oximetry decrease more than 15% under the preoperative baseline
  Interventions: Other: cerebral oximetry monitoring using INVOS™ and hemodynamic optimisation
- Blinded NIRS (Sham Comparator): Continuously monitored with cerebral oximeter but this latter is blinded to the medical team, the alarm switch off , and patients are managed with the standard care of the centre
  Interventions: Other: standard cerebral monitoring and hemodynamic optimisation

INTERVENTIONS:
Other: cerebral oximetry monitoring using INVOS™ and hemodynamic optimisation — continuous per operative cerebral oximetry monitoring associated with hemodynamic optimisation algorithm (excluding norepinephrine) if cerebral oximetry decrease more than 15% under the preoperative baseline
  Other Names: INVOS™
  Arms: open NIRS
Other: standard cerebral monitoring and hemodynamic optimisation — the patient is continously monitored with cerebral oximeter but this latter is blinded to the medical team, the alarm switch off , and patients are managed with the standard care of the centre.
  Arms: Blinded NIRS

SUMMARY:
In France, in 2007, 17 000 patients underwent carotid endarterectomy. The risk of having an ipsilateral postoperative stroke after carotid endarterectomy remains at 1-1.5%. There is no consensus concerning the best cerebral monitoring and hemodynamic optimisation during carotid cross-clamping.

The objective of this prospective, multicentric, double-blinded and randomized study is to evaluate the interest of continuous cerebral oximetry monitoring by INVOS™ cerebral oximeter to direct the hemodynamic optimisation during carotid endarterectomy and reduce the new-onset of postoperative radiological (MRI) ischemic lesions. A cost/effectiveness analysis will be conducted to estimate the impact of this monitoring versus standard care on direct and indirect postoperative costs during 120 days.

A substudy will evaluate the effect of this monitoring on neurocognitive outcome and on a serum marker of brain injury, protein S-100B

DETAILED DESCRIPTION:
After consent, patients will be randomized in two groups: one group with continuous per operative cerebral oximetry monitoring associated with hemodynamic optimisation algorithm (excluding norepinephrine) if cerebral oximetry decrease more than 15% under the preoperative baseline; the second group is continuously monitored with cerebral oximeter but this latter is blinded to the medical team, the alarm switch off , and patients are managed with the standard care of the centre.

All patients have a preoperative and a postoperative diffusion cerebral MRI to detect new onset of cerebral ischemic lesion. The amount and the volume of cerebral ischemic lesions will be scored to compare groups.

Quality of life as well as direct (medical and nonmedical) and indirect costs were collected using questionnaires during the 120 postoperative days.

A substudy including 200 patients will be conducted to compare the two groups concerning postoperative protein S-100B level and a composite score of neurocognitive tests (measured pre- and postoperatively) The trial will be conducted according to GCP

ELIGIBILITY:
Inclusion Criteria:

* Patients (male-female) over 18 y.o.
* Presenting an internal carotid stenosis requiring surgery
* Mini Mental State Examination >24 during preoperative examination
* Informed written consentExclusion Criteria:

Exclusion criteria:

* Severe renal failure or requiring dialysis
* Liver failure or cirrhosis (Child class ≥ B) or prothrombin activity<50%
* Heart failure (NYHA ≥ III), left ventricular ejection fraction < 40%, acute coronary syndrome,
* Associated surgery
* Pregnancy
* Contraindication to MRI
* History of allergy to modified gelatine or starch
* History of allergy to adhesive part of electrode

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 879 (Actual)
Dates: Start 2011-04; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The number of new cerebral ischemic lesions | Up to 3 days post-operative
  The number of new cerebral ischemic lesions observed on postoperative diffusion MRI

SECONDARY OUTCOMES:
Incremental cost-effectiveness ratio comparing the group monitored by cerebral oximeter and the standard care group | 4 months post-operative
Hospitalization length of stay | 4 months post-operative
Percentage of patient with Neurologic and neurocognitive postoperative disorders | 4 months post-operative
  * Percentage of patient with Spatiotemporal disorientation
  * Percentage of patient with aphasia
  * Percentage of patient with Facial paralysis
  * Percentage of patient with Limb sensory or motor deficit
  * Percentage of patient with Seizure
  * Percentage of patient with Balance disorder
Percentage of patient with Cardiovascular postoperative disorders | 4 months post-operative
  * Percentage of patient with myocardial infaction
  * Percentage of patient with atrial fibrillation or atrial flutter
  * Percentage of patient with acute left ventricle failure
  * Percentage of patient with Uncontrolled high blood pressure
Percentage of patient with Surgical events | 4 months post-operative
  * Percentage of patient with surgical site infection
  * Percentage of patient with haematoma evacuation
Postoperative quality of life (SF36, EQ5D tests) | 4 months post-operative
  SF36 score for quality of life assessment :
  * Physical quality score [Time Frame: Through study completion, 4 month postoperatively] Items from the SF36 (Short Form 36) survey
  * Mental quality score [Time Frame: Through study completion, 4 month postoperatively] Items from the SF36 (Short Form 36) survey
  EQ5D3L test for quality of life assessment :
  * Quality of life evaluated by the EQ 5D 3L questionnaire [Time Frame: 4 months postoperatively]
  * Quality of life, as evaluated by the use EQ 5D 3L auto-questionnaire
Incidence of death 4 month postoperatively | 4 months post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Yann Le Teurnier, MD, Principal Investigator — Nantes University Hospital
Locations (19):
- France (19):
  - Besancon University Hospital "Hôpital Jean Minjoz", Besançon
  - Bordeaux University Hospital "Haut Lévêque", Bordeaux
  - Bordeaux University Hospital "Hôpital Pellegrin", Bordeaux
  - Brest University Hospital "La Cavale Blanche", Brest
  - Caen University Hospital "Côte de Nacre", Caen
  - Dijon University Hospital "Le Bocage", Dijon
  - Le Mans Hospital, Le Mans
  - Hospital de Marie Lannelongue Plessis Robinson, Le Plessis-Robinson
  - Lyon University Hospital "Hôpital Edouard Herriot", Lyon
  - Marseille University Hospital "Hôpital de la Timone", Marseille
  - Nantes University Hospital, Nantes
  - "Nouvelles Cliniques Nantaises", Nantes
  - Nice University Hospital "Saint-Roch", Nice
  - "Groupe Hospitalier Saint-Joseph", Paris
  - "Hôpital Européen Georges Pompidou", Paris
  - Reims University Hospital "Robert Debré", Reims
  - Rennes University Hospital "Pontchaillou", Rennes
  - Strasbourg University Hospital, Strasbourg
  - Toulouse University Hospital, Toulouse

REFERENCES:
- [Derived] Le Teurnier Y, Rozec B, Degryse C, Levy F, Miliani Y, Godet G, Daccache G, Truc C, Steinmetz E, Ouattara A, Cholley B, Malinovsky JM, Portier D, Dupont G, Liutkus D, Viard P, Pere M, Daumas-Duport B, Magras PA, Vourc'h M; EMOCAR Study Group. Optimization of cerebral oxygenation based on regional cerebral oxygen saturation monitoring during carotid endarterectomy: a Phase III multicenter, double-blind randomized controlled trial. Anaesth Crit Care Pain Med. 2024 Aug;43(4):101388. doi: 10.1016/j.accpm.2024.101388. Epub 2024 May 4. PMID 38710323